CLINICAL TRIAL: NCT06729242
Title: Influence of Menstrual Cycle Phases on the Glycemic Control of Aerobic or HIIT Exercise in Adult Women With Type 1 Diabetes (DIABETEXX/2)
Brief Title: Influence of Menstrual Cycle Phases on the Glycemic Control of Aerobic or HIIT Exercise in Adult Women With Type 1 Diabetes
Acronym: DIABETEXX/2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Assistant Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024.228; PID2022-137723OB-C21 (Other Grant/Funding Number: AGENCIA ESTATAL DE INVESTIGACION)
Record Dates: First submitted 2024-12-03; First posted 2024-12-11 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type I; Menstruation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Six interventions will be carried out in a single group, being three aerobic sessions, two in two luteal phases and another in follicular phase, and other three session of high intensity interval exercise (HIIT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Aerobic session in luteal phase first menstruation (Experimental): The aerobic exercise session will begin with a 3 min resting period (sitting quietly on the cycle ergometer (0 W), followed by a 3 min warm-up at 40 W and a stepwise intensity increase by 20 W / min (to control for day-to-day variations in exercise response) until the 5% of Pmax from IET above PLTP1 is achieved (i.e. moderate steady state walking or low-intensity running or cycling). This target workload will be maintained for 30 min. Active and passive recovery periods of 3 min each will be the same as the incremental test. This session will be held on day 21 of first menstruation.
  Interventions: Other: Aerobic session
- Aerobic session in follicular phase first menstruation (Experimental): The aerobic exercise session will begin with a 3 min resting period (sitting quietly on the cycle ergometer (0 W), followed by a 3 min warm-up at 40 W and a stepwise intensity increase by 20 W / min (to control for day-to-day variations in exercise response) until the 5% of Pmax from IET above PLTP1 is achieved (i.e. moderate steady state walking or low-intensity running or cycling). This target workload will be maintained for 30 min. Active and passive recovery periods of 3 min each will be the same as the incremental test. This session will be held on day 3 of menstruation.
  Interventions: Other: Aerobic session
- Aerobic session in luteal phase second menstruation (Experimental): The aerobic exercise session will begin with a 3 min resting period (sitting quietly on the cycle ergometer (0 W), followed by a 3 min warm-up at 40 W and a stepwise intensity increase by 20 W / min (to control for day-to-day variations in exercise response) until the 5% of Pmax from IET above PLTP1 is achieved (i.e. moderate steady state walking or low-intensity running or cycling). This target workload will be maintained for 30 min. Active and passive recovery periods of 3 min each will be the same as the incremental test. This session will be held on day 21 of second menstruation.
  Interventions: Other: Aerobic session
- HIIT session in luteal phase first menstruation (Experimental): The HIIT exercise will consist of strength exercises with elastic bands. The session consists of two sets of exercise intervals of 20 s separated by 10 s of rest (i.e. 4 min in total) with a rest of 3 minutes between each set, performing in each interval a different exercise resisted by the elastic band. This session will be held on day 21 of first menstruation.
  Interventions: Other: HIIT session
- HIIT session in follicular phase first menstruation (Experimental): The HIIT exercise will consist of strength exercises with elastic bands. The session consists of two sets of exercise intervals of 20 s separated by 10 s of rest (i.e. 4 min in total) with a rest of 3 minutes between each set, performing in each interval a different exercise resisted by the elastic band. This session will be held on day 3 of first menstruation.
  Interventions: Other: HIIT session
- HIIT session in luteal phase second menstruation (Experimental): The HIIT exercise will consist of strength exercises with elastic bands. The session consists of two sets of exercise intervals of 20 s separated by 10 s of rest (i.e. 4 min in total) with a rest of 3 minutes between each set, performing in each interval a different exercise resisted by the elastic band. This session will be held on day 21 of second menstruation.
  Interventions: Other: HIIT session

INTERVENTIONS:
Other: Aerobic session — This session will consist of an aerobic training session performed on a cycle ergometer.
  Arms: Aerobic session in follicular phase first menstruation; Aerobic session in luteal phase first menstruation; Aerobic session in luteal phase second menstruation
Other: HIIT session — The HIIT exercise will consist of strength exercises with elastic bands.
  Arms: HIIT session in follicular phase first menstruation; HIIT session in luteal phase first menstruation; HIIT session in luteal phase second menstruation

SUMMARY:
Continuous glucose monitors, as a technology that aims to improve glycaemic control in patients with type 1 diabetes, must always adjust to changes in blood glucose levels in these patients, e.g. during sporting activities. In women, in particular, menstruation and its different phases can affect blood glucose levels in different ways. Therefore, this study aims to determine whether there is a different behaviour of blood glucose levels during aerobic or high-intensity exercise in different phases of menstruation. If so, we will try to model this behaviour and create specific guidelines in this regard in terms of physical exercise programming in women. In addition, the information derived from this study will be used to design better artificial pancreas systems that take into account the effects of the menstrual cycle in women.

ELIGIBILITY:
Inclusion Criteria:

Age between 18-45 years T1D with a diabetes duration for more than 2 years Glycated hemoglobin (HbA1c) < 8.5% (<69 mmol mol-1) Stable insulin regimen in the past 6 months with less than 20% change in total insulin daily dose Multiple daily injections or insulin pump Weekly physical activity of 90 min or more, but no practicing any sport as amateur or professional.

Exclusion Criteria:

Clinical conditions or use of medications (other than insulin) known to affect glycemic control (e.g., oral/parenteral steroids or metformin, among others).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean interstitial glucose | 24 hours pre-intervention and 24 hours post-intervention
  Mean interstitial glucose (mg/dL) will be measured using the FreeStyle3 as a continuous glucose meter during 6 hours, 12 hours, and 24 hours before and after both exercise sessions.
Glycemic variability | 24 hours pre-intervention and 24 hours post-intervention
  Glycemic variability (measured using the Coefficient of Variation-CV) will be measured using the FreeStyle3 as a continuous glucose meter during 6 hours, 12 hours, and 24 hours before and after both exercise sessions.
Time spent at each glucose range | 24 hours pre-intervention and 24 hours post-intervention
  Time spent at each glucose range [euglycemia (70-180 mg/dL) or Time in range (TIR), level 1 or mild hypoglycemia (54-70 mg/dL), level 2 or severe hypoglycemia (<54 mg/dL), level 1 hyperglycemia (180-250 mg/dL) and level 2 hyperglycemia (>250 mg/dL)] will be measured using the FreeStyle3 as a continuous glucose meter during 6 hours, 12 hours, and 24 hours before and after both exercise sessions.

SECONDARY OUTCOMES:
Oestrogens | pre-intervention
  Estradiol levels (pg/ml) will be measured through blood extractions and subsequent analysis in the laboratory.
Progesterone | Pre-intervention
  Progesterone (ng/mL) will be measured through blood extractions and subsequent analysis in the laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Select One, Spain

IPD SHARING:
Plan to Share IPD: No